CLINICAL TRIAL: NCT00674479
Title: Phase II Study of INCB018424 in Patients With Advanced Hematologic Malignancies
Brief Title: INCB018424 in Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0925; NCI-2012-01616 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome; Chronic Myelogenous Leukemia
Keywords: Advanced Hematologic Malignancies; Cancer; Blood; Bone marrow; Lymph nodes; JAK kinase inhibitor INCB018424 phosphate; Acute Myeloid Leukemia; AML; Acute Lymphocytic leukemia; ALL; Myelodysplastic Syndrome; MDS; Chronic myelogenous leukemia - Blast Crisis; CML; INCB018424
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB018424 (Experimental): The starting dose of INCB018424 will be 25 mg by mouth twice daily.
  Interventions: Drug: INCB018424

INTERVENTIONS:
Drug: INCB018424 — Starting dose: 25 mg by mouth (po) twice daily for 7 days each week for 4 weeks.

SUMMARY:
The goal of this clinical research study is to learn if ruxolitinib can help to control advanced hematological malignancies. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Ruxolitinib is designed to block the protein product of a mutated (changed) gene that may be important in cancer cell growth and survival.

Study Drug Administration:

If you are found to be eligible to take part in this study, every day of each 28-day cycle you will take ruxolitinib by mouth 2 times a day (in the morning and evening).

On Day 1 of each cycle, the morning dose of study drug should not be taken until you visit the clinic unless the doctor says differently.

If the doctor thinks it is necessary, your dose of study drug may be raised or lowered.

Study Visits:

On Day 1 of Cycle 1, the following tests and procedures will be performed:

* You will be asked to list any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs.

On Days 8, 15, and 22 of Cycle 1 (+/- 2 days), the following tests and procedures will be performed (these can be done at your local physician's office):

* Your medical history will be reviewed, including any drugs you may be taking.
* You will be asked if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs.
* Blood (about 2 tablespoons) will be drawn for routine tests.

On Day 1 of Cycles 2-4 (+/- 2 days) and then once every 3 months, the following tests and procedures will be performed:

* Your medical history will be reviewed, including any drugs you may be taking.
* You will be asked if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is necessary, blood (about 1 tablespoon) will be drawn to check the status of the disease.
* If the doctor thinks it is necessary, you will have a bone marrow biopsy/aspirate to check the status of the disease.
* During these visits, you will also be receiving your new supply of medication.

On Days 8, 15, and 22 of Cycles 2 and 3, blood (about 2 tablespoons) will be drawn for routine tests at your local doctor's office.

On Day 1 of Cycles 4, 7, and every 6th cycle after that (Cycles 13, 19, 25, and so on), you will have a bone marrow aspiration or biopsy to check the status of the disease. On Day 1 of Cycle 4, the bone marrow aspiration/biopsy will also look at the genes and chromosomes of the leukemia cells. If there is not enough information from the biopsy/aspirate, leftover blood will be used to look at this gene and chromosome information.

Every 2 weeks of Cycles 4-7, blood (about 2 tablespoons) will be drawn for routine tests.

You will be called once a month while you are on study. During this phone call you will be asked how you are doing, if you have experienced any side effects, and if you are taking the study drug at the correct dose and time. This phone call will take a few minutes. You will be sent a card in the mail to remind you about any study visits you need to complete.

Women who are able to become pregnant will have a urine pregnancy test if there is a suspicion of pregnancy. If the test is positive, they will then have a blood (about 1 teaspoon) pregnancy test.

Length of Study:

You may stay on study for as long as you are benefitting. You will be taken off study if you experience intolerable side effects or the disease gets worse.

End-of-Study Visit:

After you go off study you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* Your medical history will be reviewed, including any drugs you may be taking.
* You will be asked if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is necessary, blood (about 1 tablespoon) will be drawn to check the status of the disease.
* If the doctor thinks it is necessary, you will have a bone marrow biopsy/aspirate to check the status of the disease.
* Women who are able to become pregnant will have a urine pregnancy test. If the test is positive, they will then have a blood (about 1 teaspoon) pregnancy test.

This is an investigational study. Ruxolitinib is FDA approved and commercially available to treat myelofibrosis. Giving ruxolitinib to patients with advanced hematological malignancies is investigational.

Up to 120 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age.
2. Patients must have relapsed/refractory leukemias for which no standard therapies exist. Patients with poor-risk myelodysplasia (MDS) and chronic myelomonocytic leukemia (CMML) who failed prior therapy are also candidates for this protocol. Relapsed/refractory leukemias include acute non-lymphocytic leukemia (AML) by World Health Organization (WHO) classification (i.e. >/= 20% blasts), acute lymphocytic leukemia (ALL), or chronic myelogenous leukemia (CML) in blast crisis. Patients with CML who are resistant to at least two tyrosine kinase inhibitors and have no standard stem cell transplant option are also eligible.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. A female of childbearing potential must have a negative serum or urine pregnancy test at screening. Women of child-bearing potential must use acceptable contraceptive methods, and must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this trial. Nursing patients are excluded. Sexually active men must also use acceptable contraceptive methods for the duration of time on study.
5. Must be able and willing to give written informed consent.
6. In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least one week for noncytotoxic agents. Persistent clinically significant toxicities from prior chemotherapy must not be greater than grade 2.
7. Patients must have the following clinical laboratory values unless considered due to leukemic organ involvement: 1.) Serum creatinine less than or equal to 2.0 mg/dl. 2.) Total bilirubin less than or equal to 1.5x the upper limit of normal unless considered due to Gilbert's syndrome or hemolysis. 3.) Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 2.5x the upper limit of normal unless considered due to organ leukemic involvement (then 5x).
8. Patients with active central nervous system (CNS) disease are included and will be treated concurrently with intrathecal therapy. INCB018424 will not be administered by intrathecal route.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Active heart disease including myocardial infarction within the previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure.
3. Current treatment or treatment within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of study medication with another investigational medication or current enrollment in another investigational drug protocol (unless there is evidence of rapidly progressive disease in which case a shorter interval from last therapy may be acceptable).
4. Females who are pregnant or are currently breastfeeding.
5. Patients receiving therapy with intermediate or high dose steroids greater than the equivalent of 10 mg prednisone per day are not allowed.
6. Evidence of active hepatitis or human immunodeficiency virus (HIV) infection determined by screening laboratory test results or results within prior 3 months.
7. Any unresolved toxicity equal to or greater than Grade 2 from previous anticancer therapy, except for stable chronic toxicities not expected to resolve, such as peripheral neurotoxicity.
8. Incomplete recovery from any prior surgical procedures or had surgery within 4 weeks prior to study entry, excluding the placement of vascular access.
9. Uncontrolled intercurrent illness or any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.
10. In patients who are receiving medications known to be inhibitors or inducers of CYP3A4 every effort will be made to change these medications to acceptable alternatives. If this is not safely possible, patients will be excluded from participation in the study. If a patient is already on the study, must be started on a CYP3A4 inhibitor, and is demonstrating benefit from the study, they will be seen twice weekly in the first cycle and weekly in the subsequent cycles for toxicity evaluation and their dose will be modified in the event of a toxicity related to the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05-12 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Eghtedar A, Verstovsek S, Estrov Z, Burger J, Cortes J, Bivins C, Faderl S, Ferrajoli A, Borthakur G, George S, Scherle PA, Newton RC, Kantarjian HM, Ravandi F. Phase 2 study of the JAK kinase inhibitor ruxolitinib in patients with refractory leukemias, including postmyeloproliferative neoplasm acute myeloid leukemia. Blood. 2012 May 17;119(20):4614-8. doi: 10.1182/blood-2011-12-400051. Epub 2012 Mar 15. PMID 22422826
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 participants received study medication.
Period: Overall Study
Arm/Group | INCB018424
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INCB018424
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 35
Age, Continuous [Median (Full Range); unit: years] | 69 [21 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: "Time of Response " defined as the period of time from the date of first study drug administration until the first objective documentation of response. Clinical response is defined as Complete remission (CR) + Partial remission (PR) + CRp + Hematologic Improvement (HI). Participants in CR must be free of all symptoms related to leukemia and have an absolute neutrophil count (ANC) >/= 1x10^9/L, platelet count ./+ 100x10^9, normal marrow differential (</= 5% blasts). Partial remission (PR) is CR with 6-25% abnormal cells in the marrow or 50% decrease in marrow blasts. CRp is CR but platelet count < 100x10^9/L. HI is defined as for patients with pretreatment hemoglobin less than 11 g/dL, greater than 2 g/dL increase in hemoglobin; for RBC transfusion-dependent patients, transfusion independence.
Time Frame: Patients will be evaluated after each full cycle of therapy (28 days) for response.
Measure: Count of Participants; unit: Participants
Arm/Group | INCB018424
Number analyzed (Participants) | 51
Participants | 7

2. Secondary Outcome: To Determine the Pharmacokinetics (PK) Activity
Description: Exploratory sampling will be done to determine the INCB018424 PK profile. The PK parameters of INB018424 will be summarized using descriptive statistics, and the log-transformed INCB018424 PK parameters will be compared using a 1-factor analysis of variance. The mean values of the PK parameters may be compared to historical data in healthy volunteers to determine if the INCB018424 PK profile is different between patients with hematological malignancies and healthy patients.
Time Frame: Up to 3 months
Population: INCB018424 PK profile was not done because there was no historical data to compare it to. Data for this Outcome were not collected.
Arm/Group | INCB018424
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: To Determine Pharmacodynamics Activity Including the Modulation of Signal Transducer and Activator of Transcription (STAT) Protein Phosphorylation.
Description: The PD parameters will be calculated to explore preliminary evidence of PD activity by assessing the effect of INCB018424 on pre- and post-dose. If the p-STAT3/5 signaling data are sufficiently robust, an exploratory PK/PD analysis will be performed.
Time Frame: Up to 3 months
Population: The lab data was not collected so the analysis could not be done.
Arm/Group | INCB018424
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants will be assessed for adverse events from the first dose of study medication to the completion of study treatment, up to 5 years.
Arm/Group | INCB018424
All-Cause Mortality (participants affected / at risk) | 7/51
Serious Adverse Events (participants affected / at risk) | 20/51
Other Adverse Events (participants affected / at risk) | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCB018424 (N=51)
Cerebrovascular Accident (Cardiac disorders) | 1 (1)
Death (General disorders) | 6 (6)
Neutropenic Fever (Infections and infestations) | 4 (5)
Fever (General disorders) | 2 (3)
Left Basilic Vein Thrombus (Vascular disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Hemorrhage CNS (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Fall (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 2 (2)
Joint-Effusion (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-10-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT00674479/Prot_SAP_000.pdf